CLINICAL TRIAL: NCT07247968
Title: Clinical and Mechanistic Study of Subanesthetic-dose Esketamine in Modified Electroconvulsive Therapy for Adolescents With Severe Depression
Brief Title: Subanesthetic Esketamine in Modified ECT for Severe Depression in Adolescents: Clinical and Mechanistic Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Min Su (Other)
Responsible Party: Sponsor-Investigator, Min Su, Professor of Anesthesiology, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Esketamine2025-629-01
Record Dates: First submitted 2025-09-24; First posted 2025-11-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Esketamine; ECT; Depression; Adolescent
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Esketamine injection group (0.25mg/kg) (Experimental): The main anesthesiologist standing on the right side of the patient gave successive injections of esketamine (0.25 mg/kg), and 1 minute later, injected propofol (1.5mg/kg) for 30 s.After the loss of consciousness, all patients were administered 1 mg/kg of succinylcholine chloride and manually ventilated with a face mask until they regained full consciousness.
  Interventions: Drug: Esketamine injection group (0.25 mg/kg)
- Saline injection group(Consistent with esketamine injection volume) (Sham Comparator): The main anesthesiologist standing on the right side of the patient gave successive injections of saline (Consistent with esketamine injection volume), and 1 minute later, injected 1.5mg/kg of propofol in 30s.After the loss of consciousness,all patients were administered 1 mg/kg of succinylcholine chloride and manually ventilated with a face mask until they regained full consciousness.
  Interventions: Other: Saline injection group (Consistent with esketamine injection volume)

INTERVENTIONS:
Drug: Esketamine injection group (0.25 mg/kg) — The main anesthesiologist standing on the right side of the patient injects esketamine (0.25 mg/kg) sequentially, and then propofol (1.5 mg/kg) is injected 1 minute later for 30 s.After the loss of consciousness,all patients were administered 1 mg/kg of succinylcholine chloride and manually ventilated with a face mask until they regained full consciousness.
  Arms: Esketamine injection group (0.25mg/kg)
Other: Saline injection group (Consistent with esketamine injection volume) — The main anesthesiologist standing on the right side of the patient injects saline (Consistent with esketamine injection volume) sequentially, and then propofol (1.5 mg/kg) is injected 1 minute later, the injection time is 30s.After the loss of consciousness,all patients were administered 1 mg/kg of succinylcholine chloride and manually ventilated with a face mask until they regained full consciousness.
  Arms: Saline injection group(Consistent with esketamine injection volume)

SUMMARY:
The study design was a randomized, double blind, parallel controlled trial.The goal of this clinical trial is to learn if esketamine-assisted modified electroconvulsive therapy (ESK-MECT) works to treat severe depression in adolescents. It will also learn about the safety of ESK-MECT.

The sample size was calculated based on the response rate of patients with depression undergoing electroconvulsive therapy(ECT).According to the results of the pilot study,the efficacy rate of subjects receiving adjunctive esketamine was approximately 78%,while the efficacy rate of those receiving only propofol was 63%.The expected superiority difference in remission rates between the two groups was 15%(one-sided)for the power calculation.Assuming a significance level of α=0.05 and a test power of β=0.2,with a 1:1 ratio of sample sizes between the two groups,the total sample size was calculated to be 198 using the PASS software(PASS 2023).Considering a dropout rate of 10%,a total of 220 subjects were required,with 110 subjects in each group.

1. experimental group The patients were given intravenous injection of 0.25 mg / kg esketamine, 1.5 mg / kg propofol and 1 mg / kg succinylcholine in turn. After anesthesia, the patients were given electroconvulsive therapy.
2. In the control group The patients were given normal saline consistent with esketamine injection volume, 1.5mg/kg of propofol and 1mg / kg of succinylcholine. After anesthesia, the patients were given electroconvulsive therapy.

Efficacy evaluation 1. Main efficacy indicators Response rate of depressive symptoms after MECT treatment Response is defined as two consecutive HAMD-24 scores ≤ 50% before treatment after receiving MECT treatment. The response rate is calculated as the number of patients who achieved as response divided by the total number of patients receiving MECT.In this study, the 24-item version of HAMD was utilized.

Participants will:

Be randomly assigned to the esketamine group or the control group, and receive standard MECT treatment.

Have seizure parameters, seizure duration, vital signs, and complications recorded.

Complete psychiatric scale assessments, including HAMD-24, BSS, PANSS, WMS-RC and MoCA.

Be assessed at the following time points: HAMD-24 and BSS after each treatment; PANSS after each treatment course;WMS-RC and MoCA before MECT and after one treatment course.

All subjects did not discontinue antidepressants before modified electroconvulsive therapy(MECT),and they were fasting for 8 hours and no fluids for 2 hours.Three minutes before MECT,continuous qCON monitoring(Apollo-9000A,Chongqing Xideer Medical Equipment Co.,Ltd.,China)was initiated,while monitoring blood pressure,heart rate,and peripheral capillary oxygen saturation.Preoxygenation was administered for 3 minutes.The qCON monitor uses three electrodes on the forehead to collect raw electroencephalogram(EEG)signals.The qCON monitoring includes the qCON index,qNOX index,burst suppression(BS),and signal quality index(SQI).

ELIGIBILITY:
Inclusion Criteria:

* Inpatients diagnosed with Major Depressive Disorder according to the International Classification of Diseases,11th Revision(ICD-11),and scheduled for Modified Electroconvulsive Therapy(MECT);
* Aged 13 to 17 years,regardless of gender;
* Educational attainment of primary school or higher;
* Normal hearing and vision,including color perception;
* Voluntary participation in the study with signed informed consent;
* American Society of Anesthesiologists(ASA)physical status classification I-II.

Exclusion Criteria:

* Severe cardiovascular disease,significant arrhythmias,or other cardiac conditions;
* Inability to complete the assessment scales;
* History of substance abuse;
* Received electroconvulsive therapy(ECT)within 6 months prior to the study;
* Severe cerebrovascular disease,severe hypertension,intracranial hypertension,or presence of intracranial electrodes;
* Severe allergy or contraindication to propofol or succinylcholine;
* Comorbid with other psychiatric disorders.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Treatment response rate | immediately after the end of each MECT procedure
  Response is defined as two consecutive HAMD-24 scores ≤ 50% before treatment after receiving MECT treatment. The response rate is calculated as the number of patients who achieved as response divided by the total number of patients receiving MECT.In this study, the 24-item version of HAMD was utilized.

SECONDARY OUTCOMES:
Remission rate of depressive symptoms after MECT treatment | immediately after the end of each MECT procedure
  Remission is defined as a sustained HAMD scores below 10 points for two consecutive times. In this study, the 24-item version of HAMD was utilized.The remission rate is calculated as the number of patients who achieved remission divided by the total number of patients receiving MECT.
Changes in cognitive function | Immediately after the end of MECT course
  Cognitive function changes were evaluated using the Montreal Cognitive Assessment (MoCA) scales before MECT and at the end of MECT course.
The remission rate of suicidal ideation | through treatment completion, an average of 18 days
  Suicidal ideation were evaluated using the the Beck Scale for Suicidal Ideation.The remission rate of SI is calculated as the number of patients with SI remission after MECT divided by the total number of patients with SI.
Changes in psychiatric symptoms | Immediately after the end of MECT course
  Changes in psychotic symptoms that accompany depression during treatment were assessed using the Positive and Negative Syndrome Scale(PANSS) after each MECT session.
Wechsler Memory Scale-Chinese-Revision | Immediately after the end of MECT course
  The Wechsler Memory Scale-Chinese-Revision(WMS-RC)was used to assess patients'learning and memory functions before and at the end of Modified Electroconvulsive Therapy(MECT).

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data(IPD)is detailed information collected from each study participant.There are several reasons why IPD might not be shared:
  * Privacy and Confidentiality Concerns
  * Personal Identifiable Information:IPD contains sensitive information like medical history and genetic data.Sharing it without safeguards can violate privacy and lead to issues like discrimination.
  * Regulatory Requirements:Laws like GDPR require strict handling of personal data.Sharing IPD without proper anonymization and consent can result in legal problems.
  * Intellectual Property and Commercial Interests
  * Research Investment:Generating IPD requires significant resources.Researchers may want to control the data to fully exploit it for further research and publications.
  * Patent and Licensing Issues:Premature sharing of IPD can affect patentability and licensing agreements.
  * Data Integrity and Misuse
  * Quality Control:Shared IPD can be misinterpreted by others who lack context,leading